CLINICAL TRIAL: NCT04127370
Title: The Role of Bariatric Surgeries in Management of Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abo Bakr Ahmed Mahmoud, specialist( M. Sc)in Gastroenterology and Infectious Diseases Faculty of Medicine, Assiut University, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bariatric Surgery in NAFLD
Record Dates: First submitted 2019-10-01; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: NAFLD; Bariatric Surgery Candidate
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese Patients With NAFALD Undergoing Bariatric Surgeries (Experimental)
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — The Role of Bariatric Surgeries in Management of Nonalcoholic Fatty Liver Disease

SUMMARY:
The Role of Bariatric Surgeries in Management of Nonalcoholic Fatty Liver Disease

DETAILED DESCRIPTION:
The overall global prevalence of Nonalcoholic Fatty Liver Disease diagnosed by imaging is around 25.24%. The highest prevalence of NAFLD is reported from the Middle East 31.79% and South America 30.45% whereas the lowest prevalence rate is reported from Africa 13.48%.

Unlike NAFLD, Nonalcoholic steatohepatitis is more aggressive and is associated with a risk of approximately 10 to 29% of progression to cirrhosis within10 years. Therefore, early-stage NASH represents a group of patients that is most likely to benefit from treatments in order to prevent progression to cirrhosis and its complications. Obesity is the most common and well documented risk factor for NAFLD, the majority (>95%) of patients with severe obesity undergoing bariatric surgery will have NAFLD. To date, weight loss achieved via lifestyle intervention remains the mainstay of treatment of NASH.

Bariatric surgery contributes to weight loss in two main ways: restrictive procedures and malabsorptive procedures.

In 2018, the AASLD board stated that it is premature to consider foregut bariatric surgery as an established option to specifically treat NASH. Accordingly, the effects of bariatric surgery on hepatic fibrosis are still unclear. In Egypt there is lack in such type of study thus this research will conducted to evaluate the prevalence of NAFLD and NASH in obese patients undergoing bariatric surgery and to assess the role of bariatric surgery in management of NAFLD related hepatic morbidity in our locality.

ELIGIBILITY:
Inclusion Criteria:

1. Above 20 years of age
2. morbid obesity
3. severe obesity with as arterial hypertension or type 2 diabetes mellitus (T2DM),

Exclusion Criteria:

* 1- chronic liver diseases 2-Long term consumption of hepatotoxic drugs. 3-Active alcohol abuse 4-Medical or psychological contraindications for bariatric Surgery. 5-Refusal of giving a consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
change in the degree of steatosis by The Controlled Attenuation Parameter Score | one year
  change in the degree of steatosis of NAFLD patient Post Bariatric Surgery by CAP Score The Controlled Attenuation Parameter;( CAP™) This is a quantitative measurement expressed in dB/m. It varies continuously between 150 and 400 dB/m. A healthy liver will produce a measurement around 150-200, whilst a fatty liver will be measured at around 300-400 dB/m.
  CAP Score ----Steatosis Grade ------Amount of Liver with Fatty Change
  238 to 260 dB/m --S1 ----11 to 33%
  260 to 290 dB/m---- ---S2 -------34 to 66%
  Higher than 290 dB/m ----S3 ---67% or more
change in the degree of Fibrosis by Transient elastography (TE), change in the degree of Fibrosis by Transient elastography (TE), of NAFALD Patients after Bariatric Surgery NAFLD fibrosis(NFS) score and FIB-4 score. | one year
  FibroScan® is a non-invasive device that assesses the 'hardness' (or stiffness) of the liver via the technique of transient elastography FibroScan® results range from 2.5 kPa to 75 kPa
  * Fibrosis score F0 to F1: No liver scarring or mild liver scarring
  * Fibrosis score F2: Moderate liver scarring
  * Fibrosis score F3: Severe liver scarring
  * Fibrosis score F4: Advanced liver scarring (cirrhosis) Assessment of liver fibrosis by TE in NAFLD is shown in table (1) F0 to F1- F2- F3 -F4
    2 to 7 kPa 7.5 to 10 kPa
    10 to 14 kPa 14 kPa or higher ,respectively
change in the degree of Fibrosis by NAFLD fibrosis(NFS) score | one year
  change in the degree of Fibrosis by NAFLD fibrosis(NFS) score The NFS is calculated based on six readily available parameters (age, BMI, hyperglycemia, platelet count, albumin, and AST/ALT ratio) The NFS is then divided into three groups: < 1.455 which represent F0-F2, between 1.455 and 0.675 represent indeterminate, and > 0.675 represent F3-F4.
change in the degree of Fibrosis by FIB-4 score | one year
  change in the degree of Fibrosis by FIB-4 score FIB-4 index uses a combination of age, AST, ALT, and platelet count and offers dual cut-off values score < 1.45 represent unlikely advanced fibrosis and score > 3.25 represent likely advanced fibrosis, respectively
Pathological change by liver biopsy | one year
  pre and post operative liver biopsy will be taken to assess the degree of liver steatosis,inflammation and fibrosis Histological re-evaluation will be planned approximately 1 year after surgery for patient with steatohepatitis only(NAS score>3) , The histological variables will be investigated by a single specialized hepatopathologist and will be scored according to the NAFLD Activity Score (NAS recently published by the Pathology Committee of the NASH Clinical Research Network) The NAS score represents the sum of scores for steatosis (0-3), ballooning (0-2), and lobular inflammation (0-3). The score ranges from 0 to 8 with the NAS score of 5-8 considered diagnostic of NASH, the NAS score of 3-4 considered borderline NASH, and the NAS score of 0-2 considered not diagnostic of NASH. Additionally, there is a separate fibrosis stage ranging from 0 to 4 (0: no fibrosis, 1: perisinusoidal or periportal, 2: perisinusoidal and portal/periportal, 3: bridging fibrosis, 4: cirrhosis).

REFERENCES:
- [Background] Di Palma A, Alhabdan S, Maeda A, Mattu F, Chetty R, Serra S, Quereshy F, Jackson T, Okrainec A. Unexpected histopathological findings after sleeve gastrectomy. Surg Endosc. 2020 May;34(5):2158-2163. doi: 10.1007/s00464-019-07002-7. Epub 2019 Sep 11. PMID 31512035
- [Background] Papasavas P, Seip RL, Stone A, Staff I, McLaughlin T, Tishler D. Robot-assisted sleeve gastrectomy and Roux-en-y gastric bypass: results from the metabolic and bariatric surgery accreditation and quality improvement program data registry. Surg Obes Relat Dis. 2019 Aug;15(8):1281-1290. doi: 10.1016/j.soard.2019.04.003. Epub 2019 Apr 13. PMID 31477248